CLINICAL TRIAL: NCT01733758
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Monotherapy Study to Determine the Efficacy and Safety of 2 Dose Levels of Albiglutide in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Monotherapy Study to Evaluate the Efficacy and Safety of 2 Dose Levels of Albiglutide in Japanese Subjects With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113121
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Results first posted 2015-05-18 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: albiglutide; Japanese; GSK716155; Type 2 diabetes mellitus; glucagon-like peptide 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Albiglutide 30 mg weekly (Experimental): Subjects will be randomly assigned to double blind albiglutide 30 mg weekly treatment for 52 weeks
  Interventions: Drug: Albiglutide 30 mg weekly; Drug: Placebo
- Albiglutide 50 mg weekly (Experimental): Subjects will be randomly assigned to double blind albiglutide 50 mg weekly until Week 52
  Interventions: Drug: Albiglutide 50 mg weekly
- Placebo (Placebo Comparator): Subjects will be randomly assigned to double blind matching albiglutide placebo administered weekly. Subjects will then cross-over to double-blind treatment with albiglutide 30 mg weekly at Week 24 until Week 52
  Interventions: Drug: Placebo
- Liraglutide 0.9 mg daily (Active Comparator): Subjects will be randomly assigned to open-label liraglutide for 52 weeks
  Interventions: Drug: Liraglutide 0.9 mg daily

INTERVENTIONS:
Drug: Albiglutide 30 mg weekly — Albiglutide will be available as a pen injector that delivers 30mg of albiglutide
  Arms: Albiglutide 30 mg weekly
Drug: Albiglutide 50 mg weekly — Albiglutide will be available as a pen injector that delivers 50mg of albiglutide
  Arms: Albiglutide 50 mg weekly
Drug: Placebo — Albiglutide matching placebo will be available as a pen injector
  Arms: Albiglutide 30 mg weekly; Placebo
Drug: Liraglutide 0.9 mg daily — Liraglutide will be available as prefilled multidose pens that can deliver 0.9 mg dose
  Arms: Liraglutide 0.9 mg daily

SUMMARY:
This study is designed to examine the efficacy and safety of 2 dose levels of weekly subcutaneously injected albiglutide compared with placebo and an open label reference arm of daily subcutaneous injections of liraglutide, in Japanese subjects with Type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosis of Type 2 Diabetes Mellitus, treated with diet and exercise or a stable dose of 1 OAD at screening
* Body mass index (BMI) 17 to 40 kg/ m^2 inclusive
* Subjects who are OAD naïve, HbA1c between 7.0% and 10.0% at Screening and at Visit 2; for subjects who enter the study with 1 OAD, HbA1c between 6.5% and 9.5% at Screening and HbA1c between 7.0% and 10.0% at Visit 2
* Creatinine clearance >30 mL/min (calculated using the Cockcroft-Gault formula)

Exclusion Criteria:

* History of type 1 diabetes mellitus •Female subject is pregnant, lactating, or <6 weeks postpartum•
* Clinically significant cardiovascular and/or cerebrovascular disease
* Current ongoing symptomatic biliary disease, clinical signs or symptoms of pancreatitis, or a history of chronic or acute pancreatitis, as determined by the investigator
* Serum amylase >=3 ×ULN and/or serum lipase >=2 × ULN and/or subject is experiencing any symptoms possibly related to pancreatitis
* Prior use of a TZD or GLP-1R agonist within 4 months before Screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (27):
- Japan (27):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 113121 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113121 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113121 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113121 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113121 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113121 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113121 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 494 participants (par.) were randomized to one of the four treatment groups - placebo (switched to albiglutide 30 mg at Week 24), albiglutide 30 mg, albiglutide 50 mg, liraglutide (open label), 490 par. took at least one dose of study drug (Safety Population). All 490 par. were included in Intent-to-Treat Population.
Groups:
- Placebo: Participants received double-blind matching albiglutide placebo as a subcutaneous injection weekly to Week 24. After Week 24, participants received albiglutide 30 milligrams (mg) as a subcutaneous injection weekly to Week 52.
- Albiglutide 30 mg Weekly: Participants received double-blind albiglutide 30 mg as a subcutaneous injection weekly to Week 52.
- Albiglutide 50 mg Weekly: Participants received double-blind albiglutide 30 mg as a subcutaneous injection weekly until Week 4. Starting at Week 4, participants received albiglutide 50 mg as a subcutaneous injection weekly to Week 52.
- Open Label Liraglutide 0.9 mg Daily: Participants received open-label liraglutide as a subcutaneous injection daily at a dose of 0.3 mg with weekly forced uptitrations to a dose of 0.6 mg then a dose of 0.9 mg (maximum dose in Japan). The dose of 0.9 mg daily was given to Week 52.
Period: Overall Study
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open Label Liraglutide 0.9 mg Daily
Started | 77 | 160 | 150 | 103
Completed | 62 | 148 | 135 | 95
Not Completed | 15 | 12 | 15 | 8
Not completed — Adverse Event | 5 | 7 | 8 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 5 | 3
Not completed — Persistent Hyperglycemia | 3 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 2 | 2
Not completed — Non-compliance | 1 | 0 | 0 | 0
Not completed — Intro of New Anti-Diabetic Medication | 4 | 0 | 0 | 1
Not completed — Inv Decision, HbA1c not controlled | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the Safety Population.
Groups:
- Placebo: Participants received double blind matching albiglutide placebo as a subcutaneous injection weekly to Week 24. After Week 24, participants received albiglutide 30 mg as a subcutaneous injection weekly to Week 52.
- Albiglutide 50 mg Weekly: Participants received double blind albiglutide 30 mg as a subcutaneous injection weekly until Week 4. Starting at Week 4, participants received albiglutide 50 mg as a subcutaneous injection weekly to Week 52.
- Open Label Liraglutide 0.9 mg Daily: Participants received open label liraglutide as a subcutaneous injection daily at a dose of 0.3 mg with weekly forced uptitrations to a dose of 0.6 mg then a dose of 0.9 mg (maximum dose in Japan). The dose of 0.9 mg daily was given to Week 52.
- Total: Total of all reporting groups
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open Label Liraglutide 0.9 mg Daily | Total
Number analyzed (Participants) | 77 | 160 | 150 | 103 | 490
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (11.27) | 59.6 (9.00) | 57.7 (9.51) | 58.4 (9.72) | 58.4 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 35 | 36 | 22 | 118
  Male | 52 | 125 | 114 | 81 | 372
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 77 | 160 | 150 | 103 | 490

OUTCOME MEASURES:

1. Primary Outcome: Model-adjusted Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3 month period. The Baseline HbA1c value is defined as the last nonmissing value before the start of treatment. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. Based on analysis of covariance (ANCOVA): Change at Week 24 = treatment (placebo, albiglutide 30 mg, albiglutide 50 mg) + Baseline HbA1c + prior diabetes therapy + age category (<65 years versus ≥65 years). Participants who discontinued from study treatment before Week 24 had their last post-Baseline HbA1c carried forward for the analysis unless the value is past 14 days after the last dose of study drug. The open-label liraglutide group was a reference group and not included in the primary endpoint analysis model. Descriptive summary statistics are provided as a separate outcome measure.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat Population (Last Observation Carried Forward): all randomized participants who received at least 1 dose of study treatment and had a Baseline HbA1c assessment and at least one post-Baseline HbA1c assessment of HbA1c.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c in the blood
Groups:
- Placebo: Participants received double-blind matching albiglutide placebo as a subcutaneous injection weekly to Week 24. After Week 24, participants received albiglutide 30 mg as a subcutaneous injection weekly to Week 52.
- Albiglutide 30 mg Weekly: Participants received double blind albiglutide 30 mg as a subcutaneous injection weekly to Week 52.
- Open-Label Liraglutide 0.9 mg Daily: Participants received open-label liraglutide as a subcutaneous injection daily at a dose of 0.3 mg with weekly forced uptitrations to a dose of 0.6 mg then a dose of 0.9 mg (maximum dose in Japan). The dose of 0.9 mg daily was given to Week 52.
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open-Label Liraglutide 0.9 mg Daily
Number analyzed (Participants) | 77 | 159 | 150 | 0
Percentage of HbA1c in the blood | 0.25 (0.068) | -1.10 (0.047) | -1.30 (0.049) |
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 50 mg Weekly; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -1.55, 95% CI 2-sided [-1.72 to -1.39]
Statistical Analysis 2: Comparison: Placebo vs Albiglutide 30 mg Weekly; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -1.35, 95% CI 2-sided [-1.51 to -1.18]
Statistical Analysis 3: Comparison: Placebo vs Albiglutide 50 mg Weekly; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — The first test in a sequential testing procedure starting with albiglutide 50 mg versus placebo, and if significant at 0.05 level, followed by albiglutide 30 mg versus placebo; The p-value is from a 2-sided t-test to test whether the difference of least squares (LS) means (albiglutide 50 mg - placebo) is equal to zero
Statistical Analysis 4: Comparison: Placebo vs Albiglutide 30 mg Weekly; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — The second test in a sequential testing procedure starting with albiglutide 50 mg versus placebo, and if significant at 0.05 level, followed by albiglutide 30 mg versus placebo; The p-value is from a 2-sided t-test to test whether the difference of LS means (albiglutide 30 mg - placebo) is equal to zero

2. Primary Outcome: Mean HbA1c at Baseline, Week 24, and Change From Baseline at Week 24
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3 month period. The Baseline HbA1c value is defined as the last nonmissing value before the start of treatment. Change from Baseline was calculated as the value at Week 24 minus the value at Baseline. Participants who discontinued from study treatment before Week 24 had their last post-Baseline HbA1c value carried forward for the summary, unless the value was past 14 days after the last dose of study drug. The open-label liraglutide group was a reference group; descriptive statistics comparing albiglutide and liraglutide were exploratory endpoints.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat Population (Last Observation Carried Forward): all randomized participants who received at least 1 dose of study treatment and had a Baseline assessment and at least 1 post-Baseline assessment of HbA1c on or before Week 24 provided it was not past more than 14 days after the last dose of study drug intake.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open-Label Liraglutide 0.9 mg Daily
Number analyzed (Participants) | 77 | 159 | 150 | 103
Percentage of HbA1c in the blood
  Baseline | 8.16 (0.877) | 8.06 (0.783) | 8.15 (0.825) | 8.07 (0.787)
  Week 24 | 8.39 (1.066) | 6.98 (0.735) | 6.83 (0.659) | 6.87 (0.642)
  Change from Baseline | 0.24 (0.715) | -1.08 (0.619) | -1.32 (0.702) | -1.19 (0.636)

3. Secondary Outcome: Change From Baseline in HbA1c at Week 52
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3- month period. The Baseline HbA1c value is defined as the last non-missing value on or before the start of treatment. Change from Baseline was calculated as the value at Week 52 minus the value at Baseline.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (Observed Case) Population: all randomized participants who received at least 1 dose of study treatment and had a Baseline HbA1c assessment and at least one post-Baseline HbA1c assessment. Participants who discontinued from study treatment before Week 52 were not included in the analysis. No missing data were imputed.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open-Label Liraglutide 0.9 mg Daily
Number analyzed (Participants) | 62 | 148 | 135 | 95
Percentage of HbA1c in the blood | -1.07 (0.695) | -1.07 (0.790) | -1.34 (0.753) | -1.17 (0.776)

4. Secondary Outcome: Percentage of Participants Achieving Clinically Meaningful Levels of HbA1c (i.e., the Percentage of Participants Achieving Treatment Goal of <6.5% and <7.0%) at Week 24
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3 month period. Clinically meaningful levels of response in HbA1c are defined as <6.5% and <7.0%. Participants who discontinued the study before Week 24 had their last post-Baseline HbA1c value carried forwrad for the summary unless the value was past 14 days after the last dose of study drug.
Time Frame: Week 24
Population: Intent-to-Treat (Last Observation Carried Forward) Population: all randomized participants who received at least 1 dose of study treatment and had a Baseline HbA1c assessment and at least one post-Baseline HbA1c assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open-Label Liraglutide 0.9 mg Daily
Number analyzed (Participants) | 77 | 159 | 150 | 103
Percentage of participants
  HbA1c <6.5% at Week 24 | 1 | 31 | 47 | 29
  HbA1c <7.0% at Week 24 | 4 | 92 | 100 | 66

5. Secondary Outcome: Percentage of Participants Achieving Clinically Meaningful Levels of HbA1c (i.e., the Percentage of Participants Achieving Treatment Goal of <6.5% and <7.0%) at Week 52
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3 month period. Clinically meaningful levels of response in HbA1c are defined as <6.5% and <7.0%.
Time Frame: Week 52
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open-Label Liraglutide 0.9 mg Daily
Number analyzed (Participants) | 62 | 148 | 135 | 95
Percentage of participants
  HbA1c <6.5% at Week 52 | 14 | 44 | 53 | 27
  HbA1c <7.0% at Week 52 | 33 | 82 | 85 | 57

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: FPG is an indicator of efficacy. The Baseline FPG value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the FPG value at Week 24 minus the FPG value at Baseline. Participants who discontinued from study treatment before Week 24 had their last post-Baseline FPG observation carried forward for the summary unless the value was 14 days past the last dose of study drug.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open-Label Liraglutide 0.9 mg Daily
Number analyzed (Participants) | 77 | 159 | 150 | 103
Milligrams per deciliter (mg/dL)
  Baseline | 159.3 (37.07) | 157.1 (33.81) | 158.7 (32.82) | 157.2 (31.22)
  Week 24 | 167.0 (37.51) | 132.2 (26.09) | 128.8 (24.03) | 128.1 (23.68)
  Change from Baseline at Week 24 | 7.7 (31.77) | -24.9 (27.58) | -30.0 (27.83) | -29.1 (29.00)

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 52
Description: FPG is an indicator of efficacy. The Baseline FPG value is defined as the last non-missing value on or before the start of treatment. Change from Baseline was calculated as the FPG value at Week 52 minus the FPG value at Baseline.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (Observed Case) Population: all randomized participants who received at least 1 dose of study treatment and had a Baseline HbA1c assessment and at least one post-Baseline HbA1c assessment. Participants who discontinued from study treatment before Week 52 were not included in this analysis. No missing data were imputed.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open-Label Liraglutide 0.9 mg Daily
Number analyzed (Participants) | 62 | 147 | 135 | 95
Milligrams per deciliter (mg/dL)
  Baseline | 154.5 (35.65) | 154.7 (29.36) | 159.8 (33.52) | 157.4 (30.27)
  Week 52 | 131.7 (23.13) | 131.9 (24.14) | 126.3 (24.47) | 127.0 (20.78)
  Change from Baseline at Week 52 | -22.7 (27.38) | -22.8 (26.03) | -33.5 (31.10) | -30.4 (28.06)

8. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: The Baseline body weight value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the body weight value at Week 24 minus the value at Baseline. Participants who discontinued from the study treatment before Week 24 had their last non-missing weight carried forward for the summary, unless the value is past 14 days after the last dose of study drug.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open-Label Liraglutide 0.9 mg Daily
Number analyzed (Participants) | 77 | 159 | 150 | 103
Kilograms (kg)
  Baseline | 68.65 (12.088) | 69.46 (13.453) | 71.54 (12.907) | 72.65 (13.758)
  Week 24 | 68.15 (12.139) | 69.78 (13.793) | 71.50 (13.023) | 72.30 (13.459)
  Change from Baseline at Week 24 | -0.50 (1.700) | 0.32 (1.795) | -0.04 (1.976) | -0.34 (2.587)

9. Secondary Outcome: Change From Baseline in Body Weight at Week 52
Description: The Baseline body weight value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the body weight value at Week 52 minus the value at Baseline.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (Observed Case) Population: all randomized participants who received at least 1 dose of study treatment and had a Baseline HbA1c assessment and at least one post-Baseline HbA1c assessment. Participants who discontinued before Week 52 from study treatment were not included in the analysis. No missing data were imputed.
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open-Label Liraglutide 0.9 mg Daily
Number analyzed (Participants) | 62 | 148 | 135 | 95
Kilograms (kg)
  Baseline | 68.07 (11.978) | 70.07 (13.242) | 71.27 (12.801) | 72.43 (12.895)
  Week 52 | 68.00 (12.150) | 70.15 (13.536) | 70.96 (12.431) | 71.93 (12.564)
  Change from Baseline at Week 52 | -0.07 (2.179) | 0.08 (2.078) | -0.31 (2.382) | -0.50 (2.690)

10. Secondary Outcome: Time to Study Withdrawal Due to Hyperglycemia
Description: Participants who experienced persistent hyperglycemia after uptitration were to be withdrawn from the study. Hyperglycemia is defined as a fasting plasma glucose (FPG) ≥280 mg/dL (≥15.5 mmol/L) from ≥Week 2 to <Week 4, ≥250 mg/dL (≥13.9 mmol/L) from ≥Week 4 to <Week 12, or ≥230 mg/dL (≥12.8 mmol/L) from ≥Week 12 to <Week 52, confirmed a second evaluation within 7 days.
Time Frame: Baseline through Week 52
Population: Intent-to-Treat Population: all randomized par. who received at least 1 dose of study treatment and had a Baseline HbA1c assessment and at least one post-Baseline HbA1c assessment. Par. who did not conform to the protocol-defined criteria of persistent hyperglycemia with respect to FPG values defined above were not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open-Label Liraglutide 0.9 mg Daily
Number analyzed (Participants) | 77 | 160 | 150 | 103
Weeks | NA [NA to NA] — There were too few events of withdrawals due to hyperglycemia to calculate the median and confidence interval. | NA [NA to NA] — There were too few events of withdrawals due to hyperglycemia to calculate the median and confidence interval. | NA [NA to NA] — There were too few events of withdrawals due to hyperglycemia to calculate the median and confidence interval. | NA [NA to NA] — There were too few events of withdrawals due to hyperglycemia to calculate the median and confidence interval.

11. Secondary Outcome: Time to Study Withdrawal for Any Reason
Description: Time to withdrawal was calculated as the number of days between the date of first dose and the date of withdrawal plus 1. Time to withdrawal was summarized by visit.
Time Frame: Baseline through Week 52
Population: Intent-to-Treat Population: all randomized participants who received at least 1 dose of study treatment and had a Baseline assessment and at least one post-Baseline assessment (scheduled or unscheduled) of the primary endpoint, HbA1c.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open-Label Liraglutide 0.9 mg Daily
Number analyzed (Participants) | 77 | 160 | 150 | 103
Weeks | NA [NA to NA] — There were too few events of withdrawals for any reason to calculate the median and confidence interval. | NA [NA to NA] — There were too few events of withdrawals for any reason to calculate the median and confidence interval. | NA [NA to NA] — There were too few events of withdrawals for any reason to calculate the median and confidence interval. | NA [NA to NA] — There were too few events of withdrawals for any reason to calculate the median and confidence interval.

ADVERSE EVENTS:
Time Frame: On-therapy non-serious AEs and serious AEs (SAEs), events with an onset on or after the start date of study treatment and within 56 days after the date of the last dose of study treatment, are summarized through Week 52.
Description: The nonserious AEs and SAEs are reported for the Safety Population, comprised of all participants who received >= 1 dose of study treatment. Randomized treatment allocation was by design imbalanced in a ratio of 3:6:6:4 for placebo, albiglutide 30 mg, albiglutide 50 mg, and liraglutide. Non-serious AEs excludes hypoglycemia events.
Groups:
- Placebo - Before Switch: (Before Switch to 30 mg albiglutide) Participants received double blind matching albiglutide placebo as a subcutaneous injection weekly to Week 24.
- Placebo - After Switch: (After Switch to 30 mg algiblutide) After Week 24, participants received albiglutide 30 mg as a subcutaneous injection weekly to Week 52.
Arm/Group | Placebo - Before Switch | Placebo - After Switch | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly | Open Label Liraglutide 0.9 mg Daily
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/65 | 5/160 | 6/150 | 0/103
Other Adverse Events (participants affected / at risk) | 33/77 | 24/65 | 85/160 | 76/150 | 46/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Before Switch (N=77) | Placebo - After Switch (N=65) | Albiglutide 30 mg Weekly (N=160) | Albiglutide 50 mg Weekly (N=150) | Open Label Liraglutide 0.9 mg Daily (N=103)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Rathke's cleft cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Macular oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Before Switch (N=77) | Placebo - After Switch (N=65) | Albiglutide 30 mg Weekly (N=160) | Albiglutide 50 mg Weekly (N=150) | Open Label Liraglutide 0.9 mg Daily (N=103)
Nasopharyngitis (Infections and infestations) | 18 | 10 | 45 | 34 | 25
Constipation (Gastrointestinal disorders) | 3 | 3 | 14 | 17 | 7
Nausea (Gastrointestinal disorders) | 4 | 3 | 2 | 10 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 8 | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 2 | 8 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 8 | 4 | 3
Bronchitis (Infections and infestations) | 2 | 2 | 4 | 8 | 2
Pharyngitis (Infections and infestations) | 1 | 0 | 13 | 1 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 8 | 2 | 3
Eczema (Skin and subcutaneous tissue disorders) | 4 | 2 | 2 | 4 | 2
Injection site erythema (General disorders) | 0 | 1 | 3 | 9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.